CLINICAL TRIAL: NCT03563924
Title: Allo - Cancer - Thrombosis
Acronym: AlloTC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K171103J
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Cancer; Venous Thromboembolism
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Historical cohort: Patients with venous thromboembolism and cancer who follow traditional management of venous thromboembolism
- AlloTC cohort: Patients with venous thromboembolism and cancer who follow "AlloTC" specific management. "AlloTC" specific care path way develop a personalized care plan (PPS) and ensure the transmission of data (to all the interlocutors: patients and caregivers) at each step of the patient care path.
  Interventions: Other: Setting up a specific care path "AlloTC" for management of TVE in patients with cancer

INTERVENTIONS:
Other: Setting up a specific care path "AlloTC" for management of TVE in patients with cancer — Setting up a specific care path "AlloTC" for management of TVE in patients with cancer with a specific coordination nurse within the "AlloTC" multidisciplinary team as a privileged interlocutor for health professionals and patients with the aim of simplifying the care pathways and ensuring a hospital-city interface organized in collaboration with the attending physician, to develop and publicize tools available for patients and caregivers (information documents, patient monitoring protocols, etc.)
  Groups: AlloTC cohort

SUMMARY:
Management of venous thromboembolism (VTE) in patients with cancer is complex and require the intervention of many specialized health professionals, in hospital but also at home and during follow-up.

The AlloTC project aims to integrate the management of VTE within the multidisciplinary care pathway of the patient with cancer, in order to improve the management of VTE in patients with cancer: optimize treatments and follow-up with appropriate anticoagulants, monitor the implementation of good clinical practice, promote patient involvement and adherence.

The objective of this monocentric study is to evaluate the efficiency of the integration of the therapeutic management of VTE into a specific management of patient with cancer and to set up a specialized "AlloTC" team that coordinates this course of care.

For that purpose, the management of VTE and outcome of patients with cancer and VTE will be compared between two periods : traditional management and management with the "AlloTC" team.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer or haematological malignancies
* Venous thromboembolism diagnosis (symptomatic or not)

Exclusion Criteria:

* Life expectancy ≤ 3 months
* Inability to understand or sign consent
* Inability to read or understand the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with cancer or hematological malignancy and diagnosed with thromboembolic disease (symptomatic or non-symptomatic).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with appropriate care of venous thromboembolism | at 6 months
  Percentage of patients who received appropriate care of venous thromboembolism according to the latest International Good Clinical Practice (GCP) guidelines

SECONDARY OUTCOMES:
Percentage of patients with appropriate care of venous thromboembolism | at inclusion
  Percentage of patients who received appropriate care of venous thromboembolism according to the latest International Good Clinical Practice (GCP) guidelines
Percentage of patients with appropriate care of venous thromboembolism | at 3 months
  Percentage of patients who received appropriate care of venous thromboembolism according to the latest International Good Clinical Practice (GCP) guidelines
Number of calls from health professionals to the AlloTC team | at 6 months
Number of patients lost to follow-up | at 3 months
Number of patients lost to follow-up | at 6 months
Number of patients evaluated at multidisciplinary meeting | at 3 months
Number of patients evaluated at multidisciplinary meeting | at 6 months
Number of patients referred to the coordinating nurse in Oncology service | at 6 months
  Number of patients referred to the coordinating nurse in Oncology service to reassess the need for supportive care and involve health professionals (dietitian, social worker, psychologist)
Number of complications | at 3 months
  Recurrence of venous thromboembolism and bleeding episodes.
Number of complications | at 6 months
  Recurrence of venous thromboembolism and bleeding episodes.
Caregiver satisfaction survey concerning on the AlloTC team and care path | at inclusion
Caregiver satisfaction survey concerning on the AlloTC team and care path | at 3 months
Caregiver satisfaction survey concerning on the AlloTC team and care path | at 6 months
Number of patients under care for venous thromboembolism integrated into a personalized care plan as defined in the '' 2009-2013 Cancer Plan '' | at 3 months
Number of patients under care for venous thromboembolism integrated into a personalized care plan as defined in the '' 2009-2013 Cancer Plan '' | at 6 months
Number of patients accessing the venous thromboembolism information documents. | at 6 months
Percentage of patients who had at least 1 session of specialized therapeutic education | at 6 months
Assessment of the quality of life of the patient | at inclusion
  The quality of life of each patient will be evaluate using the quality of life scale 'EORTC QLC-30'
Assessment of the quality of life of the patient | at 3 months
  The quality of life of each patient will be evaluate using the quality of life scale 'EORTC QLC-30'
Assessment of the quality of life of the patient | at 6 months
  The quality of life of each patient will be evaluate using the quality of life scale 'EORTC QLC-30'
Patient satisfaction survey concerning the AlloTC team and care path | at inclusion
Patient satisfaction survey concerning the AlloTC team and care path | at 3 months
Patient satisfaction survey concerning the AlloTC team and care path | at 6 months
Number of hospitalizations in the AlloTC cohort | at 3 months
Number of hospitalizations in the AlloTC cohort | at 6 months
Hospitalization duration in the AlloTC cohort | at 3 months
Hospitalization duration in the AlloTC cohort | at 6 months

IPD SHARING:
Plan to Share IPD: Undecided